CLINICAL TRIAL: NCT00136071
Title: Randomised Prospective Blinded Trial Comparing Transvaginal Tension Free Vaginal Tape-Obturator (Outside-In) With Transobturator Tape-Mentor (Inside-Out) in Surgical Management of Urodynamic Stress Urinary Incontinence
Brief Title: Transvaginal Tension Free Vaginal Tape-Obturator (TVT-O) Versus Transobturator Tape-Mentor (TOT) in the Management of Urodynamic Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Collaborators: Henry Smith Grant (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: msakr99; Henry Smith Grant
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2005-05

CONDITIONS: Urinary Stress Incontinence
Keywords: Stress Urinary Incontinence,; TOT,; TVT-O
MeSH Terms: conditions — Urinary Incontinence, Stress

INTERVENTIONS:
Device: Transobturator tape-ARIS
Device: TVT-O

SUMMARY:
Urinary incontinence (involuntary leakage of urine) is an extremely common, distressing and socially disabling condition. It is known to affect up to 14 % of the adult female population in the United Kingdom. Sufferers tend to become social recluses, not wanting to socialise for fear of embarrassment and ridicule. It typically takes up to 5 years from the onset of symptoms for a patient to admit their problem, seek help and reach a specialist. Unfortunately, it is commonest in the elderly when the incidence is as high as 50% in some studies. Furthermore, this group of patients are the least likely to seek help, the least likely to receive help and up until recently the least likely to be cured of their problems.

Things are improving however, as everyone is more prepared to talk about this awful condition rather than accept it as a part of growing old. Furthermore, better treatments are becoming available which can help the old as well as the young.

Two years ago a new operation for urinary leakage was launched in the United Kingdom (UK). This is a smaller operation than those previously available and more suitable for the frail and elderly. We, the researchers at South Glasgow University Hospital, have been using this operation for 18 months with good success. Several versions however are now on the market, some much more expensive than the original, and perhaps not as good. We need to know which one is best and hence we intend to do a study to find out.

We aim to select patients with leakage to have one or the other operation and to follow the patients over several years to find out which operation is best, safest, lasts longest and is most acceptable to patients. Only then will we know which of the versions of this procedure we should be offering our patients.

DETAILED DESCRIPTION:
Randomised trial comparing TVT-O & TOT in surgical management of USI (Urodynamic Stress Incontinence):

Aim: To compare two transobturator tension free vaginal tape procedures; TVT-O Gynecare vs. TOT mentor for management of USI. This study will compare the surgical approach & tape material in both procedures [In-Out (TVT-O) Vs. the Out-In (TOT)] as regards to; Complication rates, Objective & subjective cure rates, Patient satisfaction & quality of life (QoL) changes.

Design: Randomised trial in a regional referral centre, approved by ethical committee.

Background: Transobturator tension free vaginal tape is currently the first choice mid-urethral tape procedure for surgical treatment of USI in our unit. The choice of the surgical approach and tape material; In-Out (TVT-O) vs. the Out-In (TOT) is currently taken predominately according to the surgeon preference without any solid clinical evidence to support that one approach or one tape is superior to the other.

Methods: All women undergoing transobturator tension free vaginal tape procedure in our department for pure USI, done as a primary anti-incontinence procedure and as the sole procedure at time of surgery, will be invited to participate in the study and will receive an information leaflet and will sign a consent form. All would have had failed or declined physiotherapy treatment. Procedures mainly take place in the surgery unit under general anaesthesia; those that are done in the main surgical list are due to patients' associated medical conditions or needing spinal anaesthesia or living in remote areas. Randomisation will be performed using sealed opaque envelopes. TVT-O & TOT will be done as originally described, we do not perform cough stress test routinely. All patients will receive intra-operative; prophylactic antibiotics & anti- inflammatory drugs if not contraindicated. Lidocaine 1% will be infiltrated into the needle pathway at the end of the procedure; 10mls. on each side. Satisfactory postoperative voiding - for the purpose of this study - is defined as passing at least 200mls with post-voiding residual urinary volume <100mls assessed at least twice.

Preoperative assessment would include:

* Detailed history & pelvic examination.
* Urodynamic assessment.
* Preoperative quality of life assessment will include:

  * Completion of the King's Health Questionnaire- version 7 (KHQ).
  * Incontinence Bothersome Scale.
  * Bristol Lower Urinary Tract Symptoms Questionnaire (BULTS).
  * Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12).

Operative assessment would include:

* Operative time
* Blood loss.
* Surgeon assessment of procedure difficulty using visual analogue score (VAS)
* Intra-operative complications:

  * Bladder/Urethral injury.
  * Haemorrhage (>200 mls.).
* Further procedures needed.
* Immediate postoperative assessment:

  * Postoperative pain assessment will include:

    * Patient self assessment using visual analogue score (VAS).
    * Unscheduled ward admission for postoperative pain.
* Postoperative voiding dysfunction will be defined as any deviation from satisfactory postoperative voiding described above. This will include assessment of:

  * Days of catheterization.
  * Intermittent self catheterization or permanent supra-pubic catheter.
  * Urethral dilatation.
  * Surgical release/excision of the tape.
  * Postoperative pyrexia,
  * Urinary tract infection (UTI).
  * Hospital stay (for medical reasons).

Outpatient postoperative assessment:

Patients will be reviewed at three months for:

* Urodynamic assessment.
* Completion of the King's Health Questionnaire- version 7 (KHQ).
* Completion of the Incontinence Bothersome Scale.
* Completion of the Patient Satisfaction questionnaire.
* Bristol Lower Urinary Tract Symptoms Questionnaire (BULTS).
* Complications: Tape erosions, De-novo urgency, Worsening of pre-existing urgency, long-term voiding dysfunction.

Patients will be reviewed at Six month, 12 month, 3 years & 5 years for:

* 24 hour Pad test.
* Completion of the King's Health Questionnaire- version 7 (KHQ).
* Completion of the Incontinence Bothersome Scale.
* Bristol Lower Urinary Tract Symptoms Questionnaire (BULTS).
* Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12).
* Completion of the Patient Satisfaction questionnaire.
* Complications: Tape erosions, De-novo Urgency, Worsening of pre-existing urgency, long-term voiding dysfunction.
* Further treatment needed.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing transobturator tension free vaginal tape procedure in our department for USI, whether a primary or secondary anti-incontinence procedure and as the sole procedure at time of surgery, will be invited to participate in the study and will receive information leaflet and will sign consent form.

Exclusion Criteria:

* Concomitant surgical procedure
* Non-english speakers
* Lack of consent

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230
Dates: Start 2005-05; Study Completion 2010-05

PRIMARY OUTCOMES:
Objective cure rates of stress incontinence according to urodynamics

SECONDARY OUTCOMES:
Improvement in total King's Health Questionnaire (KHQ) scores { > or = 10%}
Complication rates
Patient satisfaction rates

CONTACTS AND LOCATIONS:
Overall Officials: Ian Ramsay, MRCOG, Study Chair — Southern General Hospital; Mohamed Abdel-fattah, MRCOG, Study Director — Southern General Hospital
Locations (1):
- Southern General Hospital, Glasgow, United Kingdom